CLINICAL TRIAL: NCT00483717
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Study of the Safety, Tolerability, and Analgesic Efficacy of Ketorolac Tromethamine Administered Intranasally for the Acute Treatment of Migraine
Brief Title: Efficacy and Safety of Intranasal Ketorolac for the Acute Treatment of Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROX-2007-01
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Migraine
Keywords: Migraine; Ketorolac
MeSH Terms: conditions — Migraine Disorders | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Intranasal Placebo
  Interventions: Drug: Placebo
- Ketorolac tromethamine (Experimental): Intranasal ketorolac tromethamine
  Interventions: Drug: Ketorolac tromethamine

INTERVENTIONS:
Drug: Ketorolac tromethamine — 31.5 mg of ketorolac 2 x 100uL IN sprays (15% ketorolac tromethamine with 6% lidocaine hydrochloride)
  Arms: Ketorolac tromethamine
Drug: Placebo — Intranasal (IN) placebo
  Arms: Placebo

SUMMARY:
The study evaluates the efficacy and safety of using ketorolac as a nasal spray for the acute treatment of migraine.

DETAILED DESCRIPTION:
Evaluates the efficacy and safety of using ketorolac as a nasal spray for the acute treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine with or without aura (IHS criteria 1.1 and 1.2.1);
* Onset of migraine prior to age 50;
* 2-8 moderate to severe migraine headaches per month

Exclusion Criteria:

* Subjects receiving any investigational drug within 30 days before study entry;
* More than 15 headache days per month;
* Known allergy or hypersensitivity to ketorolac and/or excipients;
* Allergy to aspirin or other NSAIDs;
* Currently receiving other NSAIDs or aspirin;
* Medical history that would preclude NSAID use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Whiting, Ph D, Study Chair — American Regent, Inc.
Locations (1):
- Volker Pfaffenrath, Munich, Bavaria, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 months and 3 weeks; Medical Centers and Hospitals
Groups:
- Ketorolac Tromethamine: Intranasal ketorolac tromethamine
  Ketorolac tromethamine : 31.5 mg of ketorolac 2 x 100uL IN sprays (15% ketorolac tromethamine with 6% lidocaine hydrochloride)
- Placebo: Intranasal Placebo
  Placebo : Intranasal (IN) placebo
Period: Overall Study
Arm/Group | Ketorolac Tromethamine | Placebo
Started | 87 | 86
Completed | 63 | 65
Not Completed | 24 | 21
Not completed — Protocol Violation | 5 | 7
Not completed — Time of dosing missing | 1 | 1
Not completed — No treatment for migraine | 16 | 13
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac Tromethamine | Placebo | Total
Number analyzed (Participants) | 87 | 86 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 87 | 84 | 171
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (11.4) | 38.5 (11.6) | 38.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 76 | 158
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  Germany | 50 | 48 | 98
  Finland | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: The Number of Treated Subjects Who Became Pain-free (International Headache Society Grade of 0 = no Pain) by Observation Time Point.
Description: Pain was evaluated using a 4-point International Headache Society (IHS) scale where grade 0 = no pain, 1 = mild pain, 2 = moderate pain, 3 = severe pain
Time Frame: 2 hours after dosing
Population: Modified ITT
Measure: Number; unit: participants
Arm/Group | Ketorolac Tromethamine | Placebo
Number analyzed (Participants) | 68 | 72
participants | 12 | 7

2. Secondary Outcome: The Number of Treated Subjects Who Became Pain-free (IHS Grade 0) by Observation Time Point
Description: as for outcome 1
Time Frame: 0.5 hours post-dosing
Population: Modified ITT
Measure: Number; unit: participants
Arm/Group | Ketorolac Tromethamine | Placebo
Number analyzed (Participants) | 68 | 72
participants | 2 | 1

3. Secondary Outcome: The Number of Treated Subjects Who Became Pain-free (IHS Grade 0) by Observation Time Point
Description: as for outcome 1
Time Frame: 1 hour post-dosing
Population: Modified ITT
Measure: Number; unit: participants
Arm/Group | Ketorolac Tromethamine | Placebo
Number analyzed (Participants) | 68 | 72
participants | 12 | 4

4. Secondary Outcome: The Number of Treated Subjects Who Became Pain-free (IHS Grade 0) by Observation Time Point
Description: as for outcome 1
Time Frame: 1.5 hours post-dosing
Population: Modified ITT
Measure: Number; unit: participants
Arm/Group | Ketorolac Tromethamine | Placebo
Number analyzed (Participants) | 68 | 72
participants | 19 | 6

5. Secondary Outcome: The Number of Treated Subjects Who Became Pain-free (IHS Grade 0) by Observation Time Point
Description: as for outcome 1
Time Frame: 3 hours post-dosing
Population: Modified ITT
Measure: Number; unit: participants
Arm/Group | Ketorolac Tromethamine | Placebo
Number analyzed (Participants) | 67 | 72
participants | 22 | 10

6. Secondary Outcome: The Number of Treated Subjects Who Became Pain-free (IHS Grade 0) by Observation Time Point
Description: as for outcome 1
Time Frame: 4 hours post-dosing
Population: Modified ITT
Measure: Number; unit: participants
Arm/Group | Ketorolac Tromethamine | Placebo
Number analyzed (Participants) | 67 | 72
participants | 25 | 11

7. Secondary Outcome: The Number of Treated Subjects Who Became Pain-free (IHS Grade 0) by Observation Time Point
Description: as for outcome 1
Time Frame: 24 hours post-dosing
Population: Modified ITT
Measure: Number; unit: participants
Arm/Group | Ketorolac Tromethamine | Placebo
Number analyzed (Participants) | 67 | 72
participants | 37 | 18

8. Secondary Outcome: The Number of Treated Subjects Who Became Pain-free (IHS Grade 0) by Observation Time Point
Description: as for outcome 1
Time Frame: 48 hours post-dosing
Population: Modified ITT
Measure: Number; unit: participants
Arm/Group | Ketorolac Tromethamine | Placebo
Number analyzed (Participants) | 67 | 72
participants | 33 | 15

ADVERSE EVENTS:
Time Frame: 5 months and 3 weeks
Description: ITT population
Arm/Group | Ketorolac Tromethamine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/69 | 0/73
Other Adverse Events (participants affected / at risk) | 53/69 | 40/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac Tromethamine (N=69) | Placebo (N=73)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac Tromethamine (N=69) | Placebo (N=73)
Hypoaesthesia oral (Gastrointestinal disorders) | 5 (5) | 5 (5)
Fatigue (General disorders) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 4 (4)
Intranasal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 14 (14)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 2 (2)
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No